CLINICAL TRIAL: NCT02346799
Title: Creating Exercise Habits Through Incentives for Routines
Acronym: Routines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); National Bureau of Economic Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 821291
Record Dates: First submitted 2015-01-05; First posted 2015-01-27 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Experimental): Participants in the control group will not receive any additional treatment, apart from receiving daily emails 15 minutes before the start of their self-reported workout window. This is to control for reminder effects that may be present in the other treatment conditions. Participants in this condition will also receive a lump payment upon completion of an exit survey at the end of the intervention to equalize overall compensation.
  Interventions: Behavioral: Workout Window Reminders; Behavioral: Lump Incentive Payments
- Flexible Incentive (Experimental): Participants in the flexible incentive condition will be paid $3 or $7 for each workout they complete during the treatment period (with a limit of one incentivized workout per day, and twelve incentivized workouts during the four-week treatment period). These participants will receive daily emails 15 minutes before the start of their self-reported workout window, but they can work out anytime of the day and still receive their incentive payment.
  Interventions: Behavioral: Workout Window Reminders; Behavioral: Individual Workout Incentive Payment
- Routine Incentive (Experimental): Participants assigned to the routine incentive condition will receive the same treatment as those in the flexible incentive condition except that, in order to receive their incentive payment, they must begin their workout within their two-hour workout window. For instance, if an employee chooses a 2pm to 4pm workout window, she will receive a reminder to exercise at 1:45 pm and must swipe into the gym between 2pm and 4pm in order to receive the $3 or $7 incentive payment.
  Interventions: Behavioral: Workout Window Reminders; Behavioral: Individual Workout Incentive Payment
- Social Routine Incentive (Experimental): Participants assigned to this condition will have an identical experience to those in the routine incentive except that both partners who sign up for the study will be required to coordinate and select a common workout window. Thus, both partners will receive their daily reminders at the same time (and will be incentivized for working out at the same time). The incentive payment, however, will not be linked to whether or not a participant's partner completes a workout - only to the participant's own exercise decision.
  Interventions: Behavioral: Workout Window Reminders; Behavioral: Individual Workout Incentive Payment; Behavioral: Partner Assignment
- Holdout Control (No Intervention): If experimental enrollment exceeds target, exercise data will be collected for these additional participants, but they will receive no intervention of any kind.

INTERVENTIONS:
Behavioral: Workout Window Reminders — Participants will receive emails at prespecified times reminding them to exercise, either during a specific two hour window or at any time during the day.
  Arms: Control; Flexible Incentive; Routine Incentive; Social Routine Incentive
Behavioral: Individual Workout Incentive Payment — Participants will be paid $3 or $7 for each workout completed during the appropriate times.
  Arms: Flexible Incentive; Routine Incentive; Social Routine Incentive
Behavioral: Lump Incentive Payments — Participants will receive $20 payments for completing post treatment survey.
  Arms: Control
Behavioral: Partner Assignment — Participants will be required to have same "workout window" as partners.
  Arms: Social Routine Incentive

SUMMARY:
The purpose of this study is to determine whether healthy habits can be formed more effectively when people are rewarded for repeated engagement in a given healthy behavior at a specific, routinized time each day rather than at any time.

DETAILED DESCRIPTION:
The investigators seek to examine the effect of incentives for routine exercise on the development of persistent exercise habits. Specifically, the purpose of this study is to determine whether healthy habits can be formed more effectively when people are rewarded for repeated engagement in a given healthy behavior at a specific, routinized time each day rather than at any time. Through a partnership with a Fortune-500 company, the investigators plan to run a large-scale, randomized field controlled trial with approximately 3,000-4,000 participants aimed at increasing exercise rates (as measured by gym visits). During an incentivized four week intervention period, the investigators will encourage participants to select a two-hour window during the day when they feel they are most willing and able to exercise. Depending on condition, participants will [a] receive no further instruction or incentives (control condition), [b] receive a $3 or $7 bonus for each day they exercise during the incentive period (flexible incentive condition), or [c] receive a $3 or $7 bonus for each day they exercise if and only if they exercise within their specified "workout window" (routine incentive condition). Additionally, participants in a fourth condition, the social routine incentive condition, will face the same incentives as those in the routine incentive condition, but will be required to coordinate the workout window they select with a partner in their office. The investigators predict that the less flexible incentives will lead to greater habit formation than flexible incentives, producing larger and longer-lasting increases in exercise post-intervention. The investigators further predict that coordinating with a workout partner will produce even stronger habit formation. The investigators will collect and analyze data from participants' worksite gyms, which track gym entries and exits, as well as pedometer data when available.

Our experiment will recruit employees at a Fortune-500 company who wish to exercise more. Recruitment will be done through an email and poster campaign. The registration stage will take approximately four weeks. All employees at all offices with on-site gyms will be eligible to enroll and upon enrollment will be asked to select a partner who works in the same office and who is also enrolling. Enrolling employees will also be asked to indicate their preferred daily workout time (a two hour "workout window") and to provide basic demographic and exercise-related information (e.g., gender, age, height, weight, number of gym visits per week). If registration exceeds the target sample size (4,000 employees), priority for enrollment will be given to employees who do not already exercise regularly (at least twice a week). The remaining participants will be assigned to a "holdout control" condition. Once registration is closed, participants will be assigned randomly (at the pairs level) to one of the four experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be full-time employees of partner company

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2702 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Average weekly number of 30+ minute visits to company gym | Up to one year
  Number of times per week participants enter the company gym and exit at least 30 minutes later
Duration of habit | Up to one year
  Length of time that weekly gym visits takes to return to baseline level

SECONDARY OUTCOMES:
Activity level as measured by Fitbit pedometers | Up to one year
  Number of steps taken during workouts, as measured by Fitbit pedometers

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States